CLINICAL TRIAL: NCT00817102
Title: Validation of Stenosis Assessment by Coronary Artery Computed Tomography Against Invasive Measurements of Fractional Flow Reserve in Patients With Significant Coronary Artery Stenoses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Piedmont Healthcare (Other)
Responsible Party: Charles Brown, MD, Piedmont Healthcare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ATLANTA II
Record Dates: First submitted 2009-01-02; First posted 2009-01-06 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Coronary Artery Stenosis
Keywords: coronary artery stenoses
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CorCTA (Other): Fractional Flow Reserve (FFR), Intravascular Ultrasound (IVUS), Virtual Histology (VH) or some combination of these three procedures
  Interventions: Procedure: FFR, IVUS, VH, or combination of the three

INTERVENTIONS:
Procedure: FFR, IVUS, VH, or combination of the three — Fractional Flow Reserve (FFR), Intravascular Ultrasound (IVUS), Virtual Histology (VH) or some combination of these three procedures will be completed during the cardiac catheterization procedure.

SUMMARY:
This study will evaluate the effectiveness of CorCTA by comparing the results of the test with another imaging method called Fractional Flow Reserve (FFR), which is done as a part of the cardiac catheterization.

DETAILED DESCRIPTION:
Invasive X-ray coronary angiography remains the "reference standard" for the evaluation of coronary artery stenoses. Recently, coronary artery computed tomography angiography (CorCTA) has been introduced as a non-invasive method for the evaluation of coronary artery stenoses and has been shown to be highly accurate in stenosis detection when compared to invasive X-ray angiography. While invasive X-ray angiography and CorCTA evaluate morphological features of coronary arterial plaques, fractional flow reserve is an invasive measure of the hemodynamic significance of a stenosis obtained in the catheterization laboratory by measuring changes in intracoronary arterial pressure before and after maximal vasodilation induced by intracoronary adenosine. An FFR value less than 0.75 has been shown to predict ischemia in vascular beds distal to the stenosis by radionuclide perfusion modalities and has been shown to be associated with worse outcomes. Therefore, FFR is considered to be an invasive hemodynamic "reference standard" for the evaluation of the hemodynamic significance of coronary arterial stenoses. While intravascular ultrasound (IVUS) can provide additional morphological information in intermediate stenoses, it can not provide further functional information and cannot be used in more significant stenoses as the IVUS probe cannot be advanced through stenotic lesions.

We are currently conducting investigation in the validation of CorCTA against FFR in intermediate coronary artery stenoses (40-70%) (see below under "Preliminary Data"). However, CorCTA has not been validated against invasive hemodynamic measurements of fractional flow reserve in patients with stenoses >70% by invasive X-ray angiography. We hypothesize that CorCTA-derived measurements are accurate in the diagnosis of hemodynamically significant coronary artery stenoses, using FFR as the reference standard in patients with coronary artery stenoses>70%.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-85
* Presence of at least one obstructive coronary artery stenosis as defined by:

  * Previous catheterization or CT angiogram with any lesion 70% or greater
  * Previous positive functional stress test (this does not include CTA alone)
* Ability and Willingness to provide informed consent
* Ability and Willingness to perform required follow up procedures

Exclusion Criteria:

* History of coronary artery bypass graft surgery
* Previously revascularized lesion
* Creatinine>1.6 mg/dL or GFR<30 pre-procedure per institutional standards
* Known Pregnancy
* Inability to perform CTA
* Arrhythmia precluding diagnostic CT examination
* Contrast agent allergy that cannot be adequately premedicated
* Severe PVD precluding cardiac catheterization
* Patient not a candidate for IVUS and FFR
* Inability or unwillingness to provide informed consent
* Inability or unwillingness to perform required follow up procedures

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-11; Primary Completion 2011-11 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The CT-derived endpoints: Study lesion %DS predicting FFR<0.75; %AS predicting FFR<0.75; MLD predicting FFR<0.75; Study lesion MLA predicting FFR<0.75; IVUS-derived endpoints: Study lesion MLD predicting FFR<0.75; MLA predicting FFR<0.75 | Upon completion of tests

CONTACTS AND LOCATIONS:
Locations (1):
- Piedmont Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Vazquez-Figueroa JG, Rinehart S, Qian Z, Joshi PH, Sharma A, Lee J, Anderson H, Murrieta L, Wilmer C, Carlson H, Taylor K, Ballard W, Karmpaliotis D, Kalynych A, Brown C 3rd, Voros S. Prospective validation that vulnerable plaque associated with major adverse outcomes have larger plaque volume, less dense calcium, and more non-calcified plaque by quantitative, three-dimensional measurements using intravascular ultrasound with radiofrequency backscatter analysis : results from the ATLANTA I Study. J Cardiovasc Transl Res. 2013 Oct;6(5):762-71. doi: 10.1007/s12265-013-9473-0. Epub 2013 May 22. PMID 23695823